CLINICAL TRIAL: NCT04098536
Title: Acute Exposure to Diesel: Prolong Effects on Inflammation and Vasculature
Acronym: DEVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Dimitris Tousoulis, Professor Dimitris Tousoulis, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 14/20/7/2016
Record Dates: First submitted 2019-09-15; First posted 2019-09-23 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Vehicle Emissions

STUDY DESIGN:
Intervention Model Description: Cross over double blind
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diesel Exposure (Experimental)
  Interventions: Behavioral: Diesel exhaust
- Filtered Air Exposure (Placebo Comparator)
  Interventions: Behavioral: Diesel exhaust

INTERVENTIONS:
Behavioral: Diesel exhaust — Exposure to diesel exhaust fumes
  Other Names: Filtered air exposure

SUMMARY:
Cross-over double-blind study. Healthy subjects will be exposed to diesel exhaust fumes and/or filtered air during a 2-hour session. Several parameters will be assesed i.e. endothelial function will be assessed with flow mediated dilation (FMD) techniques, arterial stiffness with pulse wave velocity (PWV) and reflected waves with augmentation index (AIx). C reactive protein (CRP), fibrinogen, protein C levels and protein S activity will be also measured. Heart rate variability and standard deviation of normal to normal intervals R-R intervals (SDNN) will be used to assess sympathetic activity. Measurements were assessed before, 2 and 24 hours after diesel exposure.

DETAILED DESCRIPTION:
Introduction Diesel and its products represent one of the most common pollutants affecting people living in urban and rural areas of the world. The majority of patients attending emergency departments are likely to have been subjected to chronic exposure to diesel engine exhaust fumes particularly those living in proximity to busy city roads and highways. Diesel exhaust fumes are considered to contribute to over 50% of atmospheric particles with a mass of less than 10 μM (PM10) average aerodynamic diameter, which is responsible for air pollution. For fine particle matter lower than 2.5 μM (PM2.5) and extremely small particles below 0.1 μM in diameter, the contribution to air pollution is much greater. These particles are small enough to be inhaled and deposited in the lungs where they can exert deleterious effects.

In Europe and Japan, epidemiological studies have demonstrated high rates of cardiovascular morbidity, as well as acute and chronic respiratory disease, following occupational exposure to diesel exhaust fumes. Experimental animal studies have also shown that exposure to diluted diesel engine emission impairs left ventricle systolic performance, sympathetic drive, fibrosis/fibrinolysis and accelerates atherosclerosis. Epidemiological studies and experimental animal models are, however, rather imprecise regarding the mechanisms responsible for these effects and the clinical impact of chronic diesel exhaust fumes exposure. Moreover, although a relationship has been documented between acute coronary syndromes (ACS) and acute exposure to diesel engine exhaust fumes, it is not known whether relatively short-term exposure can cause prolonged inflammatory responses and/or affect endothelial function and vessel wall properties in such a way as to potentially promote the development of atherosclerotic changes.

The purpose of this study is to assess the impact of short-term exposure to Diesel exhaust fumes on arterial elasticity, vascular function and inflammatory biomarkers.

Methods Study population Volunteers will be included in this randomized, double blind, crossover study All volunteers who qualified for study entry will be free of cardiovascular disease, hypertension, diabetes mellitus, pulmonary disease and acute inflammatory or chronic diseases. Subjects who will be found to have an abnormal baseline 12-lead electrocardiogram and/or impaired respiratory function tests will be excluded from the study.

Individuals taking cardiovascular medications, antioxidant or vitamin supplementation, oral contraceptives or anti-inflammatory agents during the two months prior to inclusion in the study will be excluded.

Women receiving hormone replacement therapy and premenopausal women with irregular menstrual cycles will also excluded from the study. All women selected for the study will underwent pregnancy tests before each study session.

Study Design This is randomized double-blind, cross-over study. All subjects will be exposed to air or pollutants in two sessions which will took place 4 weeks apart between 8.00 and 10.00 a.m. in an ad hoc laboratory. In each session, the subjects will underwent a 2-hour exposure period to controlled amounts of diesel exhaust fumes or filtered air. In each session, measurements of markers of vascular function (flow mediated dilation, pulse wave velocity and augmentation index), sympathetic activity and blood tests depicting the inflammatory and fibrinolytic profile will took place. These measurements will be performed at baseline (before exposure-T0), at the end of the 2-hour session (T2) and 24 hours after the end of exposure (T24) (Figure 1).

Measurements in each women participating in the study will be performed at the same phase of the menstrual cycle (late luteal phase). The participants will refrained from drinking alcohol or caffeinated fluids and using medications containing caffeine, or smoking. All volunteers will be assessed after having been in the fasting state for at least 8 h. Participants will instructed to avoid changes in diet and physical activity habits during the study period.

Diesel exhaust and filtered air exposure Volunteer exposure to diesel exhaust fumes will carried out on a specially designed 30m2 room which was hermetically sealed. The diesel exhaust fumes will be produced by a diesel engine (2500 cc and 100-150HP) and dispensed through a pipe system into the exposure room. Prior to study entry, indoor levels of carbon monoxide (CO) along with concentrations of fine airborne particulate matters (PM2.5) will be measured, controlled and kept within the desired limits using portable environmental instrumentation. In order to secure adequate levels of exposure to PM2.5 and CO, all measurements will be controlled and compared to the respective standards of the European Commission. Specifically, 25 µg/m3 (mean annual limit) for PM2.5 particles and 10 µg/m3 (maximum daily 8 hour mean) for CO.

Vascular measurements Endothelial function evaluation Using a linear array ultrasound (U/S) transducer endothelial function will be evaluated by estimating flow mediated dilation (FMD) in the brachial artery, as per standardized protocols.

Central arterial stiffness measurements Carotid-femoral pulse wave velocity (PWV), an index of aortic stiffness, will be calculated from measurements of pulse transit time and the distance between 2 recording sites (PWV = distance, in meters, divided by transit time, in seconds) using a well-validated non-invasive device (SphygmoCor; AtCor Medical, Sydney, Australia) as previously described.

Measurement of wave reflections The AIx of the central (aortic) pressure waveform will be calculated as a composite index of wave reflections and arterial stiffness using a validated, commercially available system (SphygmoCor; AtCor Medical, Sydney, Australia) which employs the principle of applanation tonometry. Waveforms of radial pressure will be calibrated according to sphygmomanometric systolic blood pressure and diastolic blood pressure measured in the brachial artery. Because the AIx is influenced by changes in HR, it was corrected as appropriate (corrected for a steady HR of 75 bpm; AI75).

Sympathetic activity assessment Heart rate variability (HRV) expresses the impact of the autonomic nervous system on heart activity. Low HRV may be attributed to increased sympathetic tone and has been found to be associated with increased cardiovascular morbidity and mortality. Sympathetic activity will be evaluated by calculating HRV with continuous electrocardiographic study (ECG) which was recorded for 20 minutes by a Holter device. ECG data will then transferred onto a computer for assessment of HRV, which was performed in accordance with current international guidelines, and standard deviation of normal to normal intervals (SDNN) will be measured. (Holter software, Synescope, version 3.1, ELA Medical, France).

Fibrinolysis and inflammation markers A fasting venous blood sample will collected by venipuncture at baseline (before exposure-T0), at the end of the 2 hours session (T2) and 24 hours after the end of exposure (T24). Venous blood samples will be centrifuged at 3000 rpm and serum was collected and stored at -80 C until assayed.

The prothrombotic status was assessed by measuring levels of fibrinogen using the Multifibren® U system. Fibrinolytic activity will be assessed with measurements of protein C plasma levels and protein S activity, which were measured by the STA® - Staclot® Protein C kit and HemosIL™ Protein S Activity kits, respectively. Furthermore, changes from baseline in the inflammatory profile induced by diesel exhaust fumes will be studied by measuring serum C-reactive protein (CRP) using the Architect Abbott device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Chronic diseases Cardiovascular diseases Respiratory diseases Pregnacy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Endothelial function assesment | 24 hours
  The following outcome will be evaluated
  Changes over time of :
  Flow mediated dilation (FMD) mesured in the branchial artery with ultrasound. Units %
Arterial Stifness | 24 hours
  The following outcome will be evaluated
  Changes over time of :
  Carotid-femoral pulse wave velocity (PWV), measured non invasively Units: m/sec

SECONDARY OUTCOMES:
Sympathetid Activity | 24 hours
  Change over time of Standard deviation of ECG RR intervals Units: msec
Inflammation | 24 hours
  Cgange over time of C reactive protein levels Units Mg/dl

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - 1st Cardiology Department, Hippokration General Hospital, Athens, Attica
  - Evangelos Oikonomou, Athens, Please Select

IPD SHARING:
Plan to Share IPD: Undecided